CLINICAL TRIAL: NCT02883881
Title: Correlation Between Eye Rubbing and Keratoconus Severity in a Treatment-naive Keratoconic Population
Acronym: FROTT EYES
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-02Obs-CHRMT
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- No eye rubbing
- with eye rubbing

SUMMARY:
determination if, within a keratoconic population, strong eye rubbing was correlated with visual acuity, spherical equivalent value, biomicroscopic signs, corneal pachymetry, keratometry, and tomography classification determinating keratoconus stage.

DETAILED DESCRIPTION:
A retrospective study was performed between november 2014 and october 2015 in the Metz Hospital Center. Were included 33 patients presenting with treatment-naive keratoconus. Patients responded to a questionnaire that assessed eye rubbing habits, family history of keratoconus, history of atopy. 2 groups were separated: group 1 constituted by 15 eyes with no eye rubbing, and group 2 constituted by 18 eyes with moderate or severe eye rubbing. The following informations were collected: best visual corrected acuity (BCVA), spherical equivalent value (SEV), corneal opacities or Vogt striae. For each eye were performed an anterior segment OCT (AS-OCT) to determine the OCT stage for keratoconus (Fourrier domain OCT classification, 2013), and a Scheimpflug camera imaging to determine the maximal keratometry (Kmax) and the minimal corneal thickness (MCT).

ELIGIBILITY:
Inclusion Criteria:

* patients presenting with treatment-naive keratoconus.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting with treatment-naive keratoconus.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
visual acuity | month 1